CLINICAL TRIAL: NCT03692273
Title: A Within-Scar, Randomized Control Trial Comparing Fractional Ablative Carbon Dioxide Laser to Non-Energy-Based, Mechanical Tissue Extraction and No Treatment
Brief Title: Randomized Control Trial of CO2 Laser to Treat Hypertrophic Burn Scar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jonathan Friedstat, Instructor of Surgery, Harvard Medical School, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MB170043
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Burns; Hypertrophic Scar
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: Patients will receive all three interventions (laser, 0.5mm punch biopsy, and no treatment) within their study scar.
Who Masked: Outcomes Assessor
Masking Description: The provider and patient will know which area is randomized to the three treatments. The assessors of the primary and secondary outcomes will be blinded to which treatment was provided to each of the three areas within the study scar.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Laser (Experimental): Laser treatment to 3x3cm2 area. It will receive the Luminous ultra pulse fractional ablative carbon dioxide laser at 150mJ, 3% density and 250Hz.
  Interventions: Procedure: Luminis ultrapulse fractional ablative carbon dioxide laser
- 0.5mm punch biopsy (Experimental): 0.5mm punch biopsy area. This area will receive 0.5mm punch biopsies 75 per cm2 at a depth of 5mm.
  Interventions: Procedure: 0.5mm punch biopsy
- No treatment (No Intervention): 3x3cm2 area designated as no treatment that will serve as a control

INTERVENTIONS:
Procedure: Luminis ultrapulse fractional ablative carbon dioxide laser — This laser will target water molecules and ablate columns of tissue that are approximately 3mm deep.
  Arms: Laser
Procedure: 0.5mm punch biopsy — punch biopsies will be performed to remove approximately equivalent volumes of tissue compared to the laser
  Arms: 0.5mm punch biopsy

SUMMARY:
Laser treatment of hypertrophic burn scars has become increasingly popular for improving scarring in burn survivors. Despite its common use, there a gap in knowledge regrading randomized control trials that demonstrate whether the laser is beneficial. Such a trial is important because if it shows the laser does work, it would provide the evidence to make such treatments more accessible to all patients.

Furthermore, there is no knowledge whether the burn injury used to remove tissue is beneficial or not. This study aims to evaluate the laser treatment, removal of similar tissue amounts with 0.5mm punch biopsies, to controls to fill this knowledge gap.

The hypothesis is the laser is beneficial at improving patient's burn scars. Also the punch biopsies work better at improving scars by removing tissue without burning and injuring the surrounding tissue as the laser does.

To evaluate these treatments (laser, punch biopsies, and no treatment), 3 small areas will be chosen in a study scar area that meets specific criteria to receive . Patients will still be able to receive laser and burn reconstruction procedures in all other areas not involving the study scar area that are clinically indicated.

In the study, the scar will be evaluated with photographs, surveys, and tissue samples taken either while under anesthesia except for one set taken with numbing medicine. The tissue samples will be looked at under a microscope to see how the treatments change the scar tissue. The tissue will also have tests done to evaluate how the laser impacts genes from cells in the scar tissue.

Lastly, to understand how reconstructive procedures (laser and surgical treatments) change a patient's quality of life, patients will be asked a limited set of questions to learn more how these procedures improve their lives.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older
* Must be medically fit to undergo laser/reconstructive procedure
* Must have symptomatic HTBS for which they are already planning to undergo laser treatment. The symptomatic HTBSs may include the study scar area, but there must be other areas that the patient is getting treated with laser besides the study scar.
* The HTBS must have occurred from a burn injured area either treated by skin grafts or allowed to heal secondarily.
* Be willing and able to participate in the study with a year of follow-up
* Must be able to answer surveys on their own, and not rely on surrogates
* Not be pregnant or planning to become pregnant during the treatment phase of the study

Study Scar Inclusion Criteria:

* The study scar must be at least 3mm thick
* For Extremities, no surgical treatment can be performed on joint space above or below the target area

  * If the study scar is over a joint, then no surgical treatments can occur to the body part above or below it
* When the study scar is on the trunk or neck, it must not be on continuity or adjacent to any area of planned surgical treatment.
* Study Scar Size: The study scar can either be within an area of homogenous HTBS or be an area of HTBS surrounded by normal tissue if it meets the following size criteria:
* Within HTBS For treatment areas within burn scars, it must be 65cm2 or larger to permit 3 treatment areas that are 3 x 3cm with a 1cm wide segment of untreated scar between it.
* Surrounded by normal tissue For treatment areas surrounded by normal skin, the treatment area must be 33cm2 or greater, contain similar 3x3cm treatment areas, and have intervening segments of 1cm of scar between treatment areas. A border around the scar, is not required here because it is surrounded by normal skin.

Exclusion Criteria:

* Previous laser or reconstructive procedures for the treatment of their HTBS in the study scar or adjacent tissue.
* Steroids, immunosuppressive medications, chemotherapy or other medications that can delay their wound healing/immune function.
* Medical Conditions that preclude laser treatment or general anesthesia if needed
* Cognitively unable to complete PROMs on their own
* The study area should not be part of a contracture or other hypertrophic scar that would be better treated with surgical procedures.
* The study scar must not be adjacent to/in continuity with areas of HTBS that are planning to be treated with surgical interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale | 14 months (from first treatment to follow-up)
  scar scale to evaluate severity of hypertrophic burn scars This is a 3 question scale, the first question graded from 0-3, the second and third questions graded from 0-5. The final score is the sum of the scores of the three questions, giving a possible total score range of 0-13. The higher the score, the worse the outcome.

SECONDARY OUTCOMES:
photography of treatment areas in scar for evaluation | 14 months (from first treatment to follow-up)
  Evaluation of photographs of the treatment areas in the study scar
elasticity of treatment areas of scar | 14 months (from first treatment to follow-up)
  Measure elasticity using a cutometer
histology of treatment areas of scar | 14 months (from first treatment to follow-up)
  tissue samples will be evaluates for changes in cell architecture, collagen, and cells within the scar
Gene expression | 14 months (from first treatment to follow-up)
  Inflammatory gene expression will be evaluated between laser treatment and control tissue

OTHER OUTCOMES:
Patient Reported Outcome Measures Burn Specific | 14 months (from first treatment to follow-up)
  LIBRE (Life Impact Burn Recovery Evaluation)
Patient Reported Outcome Measures Generic | 14 months (from first treatment to follow-up)
  PROMIS 28 (Patient-Reported Outcomes Measurement Information System)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Friedstat, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No